CLINICAL TRIAL: NCT06260449
Title: Different Treatment Approaches of Presumed Trematode-Induced Uveitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ibrahim, Physician, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Trematode
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Uveitis
Keywords: Trematode; Pearl shape granuloma
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Intervention Model Description: Single group tested by intervention and medical treatment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgical removal (Experimental): Surgical removal of the whitish granuloma
  Interventions: Procedure: Surgical removal
- Medical treatment (No Intervention): Topical and systemic steroid
- Laser treatment (Experimental): Argon laser
  Interventions: Procedure: Surgical removal

INTERVENTIONS:
Procedure: Surgical removal — Removal of the granuloma
  Arms: Laser treatment; Surgical removal

SUMMARY:
Different Treatment Approaches of Presumed Trematode-Induced Uveitis including periocular injection and medical treatment Nd laser treatment

DETAILED DESCRIPTION:
Uveitis, characterized by inflammation of the uvea, is a complex and potentially sight-threatening ocular condition that can result from various etiologies. Among causes of uveitis, trematode-induced uveitis represents a distinct and intriguing subset characterized by the presence of a single or multiple pearl like nodules in the anterior chamber (AC) or less commonly in the conjunctive, cornea or even in the ciliary body and posterior segment. Trematodes, or parasitic flatworms, have been implicated in causing uveitis through the migration of larvae or adult worms into the eye, triggering an inflammatory response 1. Despite its rarity, trematode-induced uveitis poses diagnostic and therapeutic challenges due to the diversity of trematode species and the lack of standardized treatment protocols 2. The treatment of trematode-induced uveitis typically involves addressing the underlying parasitic infection and managing the associated inflammation. Various treatment modalities have been reported in literature. Antiparasitic medications have been tried by some authors. Advantages include targeting the underlying cause by killing the parasites. In addition, systemic medications can reach distant sites of infection However, there is no evidence that the parasite is actually living in ocular tissues and the inflammatory process may be directed against already dead parasite 3. Also, they may have side effects. Effectiveness depends on the specific type of trematode and its susceptibility to the chosen medication. Steroid Therapy is considered the gold standard treatment including topical steroids and periocular Injection of Triamcinolone) Advantages: Reduces inflammation in the eye. Provides symptomatic relief. Disadvantages: Does not address the underlying cause (parasitic infection)4. Prolonged or high-dose steroid use may lead to side effects, such as increased intraocular pressure or cataract formation. In resistant cases Surgery has been advocated by many authors Advantages: Surgical removal of nodules may be considered in specific cases. Can be beneficial in cases of severe complications, such as retinal detachment5. Disadvantages: Invasive procedure with associated risks and is mainly aimed at managing complications.

Laser Therapy has been reported to destroy the pearl like nodules using Argon laser Potential damage to surrounding healthy tissue is the main drawback.

Therefore, there is no consensus about the best line of treatment for this entity Rational for this study: Understanding the available treatment options is crucial for healthcare professionals involved in the care of patients with this condition7

ELIGIBILITY:
Inclusion Criteria:

Clinical Presentation:

Presence of Uveitis: Include patients with clinically diagnosed uveitis, characterized by inflammation of the uvea9.

Suspicion of Trematode Etiology: Include cases where there is a reasonable suspicion or evidence suggesting trematode-induced uveitis based on clinical picture of pearl like whitish AC or subconjunctival nodules characteristic for this specific entity, history of swimming in local ponds and canals in endemic areas.10

Diagnostic Confirmation:

Positive Diagnostic Findings: Include patients with characteristic clinical picture and exclusion of other causes of granulomatous uveitis by appropriate laboratory tests and imaging modalities.11

Severity of Uveitis:

Disease scores at presentation for parasitic granulomatous uveitis Parameter range score Diameter of AC lesion >3mm 1 3-5mm 2 <5mm 3 Grade of AC inflammation +.5 to+1 1

* 2 to +3 2
* 4 3 Complications at presentation none 0 Retro corneal scar or corectopia 1 Cataract 2 Glaucomatous optic atrophy 3

Eyes with scores > 5 were started on steroid therapy. Patients with severity scores <= 5at presentation were advised for surgical excision of the AC lesions.

Based on SUN grading scheme for AC cells.

Age and Gender:

All Ages: Consider including patients of all age groups. Both Genders: Include both males and females

Exclusion Criteria:

Alternative Diagnoses:

Presence of Other Ocular Diseases: Exclude patients with other causes of uveitis12.

Concomitant Systemic Infections: Exclude patients with concomitant systemic infections that may independently cause uveitis.

Patients unwilling to participate in the study

Treatment History:

Previous Treatment for Trematode-Induced Uveitis: Exclude patients who have previously undergone treatment specifically for trematode-induced uveitis13.

Non-Compliance: Exclude patients with a history of non-compliance with prescribed treatments.

Contraindications to Specific Treatments:

Contraindications to Medications: Exclude patients with known contraindications to specific antiparasitic medications or corticosteroids.

Ineligibility for Surgery: Exclude patients who are not suitable candidates for surgical interventions14.

Pregnancy and Lactation:

Pregnant or Lactating Women: Consider excluding pregnant or lactating women due to potential risks associated with certain treatments15

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2024-10-21 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Surgical removal | Baseline
  Surgical wash of granuloma with topical and systemic steroid

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amin RH, Abdullatif AM. Management of presumed trematode-induced granulomatous intermediate uveitis. Eye (Lond). 2023 Aug;37(11):2299-2304. doi: 10.1038/s41433-022-02336-4. Epub 2022 Dec 7. PMID 36477731
- [Background] El Hefny E, Sabry D, Sewelam A, El Nokrashy A. Characteristics of Childhood Presumed Trematode-Induced Granulomatous Anterior Uveitis Using Ultrasound Biomicroscopy. Ocul Immunol Inflamm. 2022 Oct-Nov;30(7-8):1604-1608. doi: 10.1080/09273948.2021.1922709. Epub 2021 May 20. PMID 34014799
- [Background] Amin RM, Radwan AE, Goweida MB, El Goweini HF, Bedda AM, Lotfy WM, Ahmed ARH. Management of presumed trematode induced granulomatous uveitis in pediatric patients. Jpn J Ophthalmol. 2019 Jan;63(1):119-125. doi: 10.1007/s10384-018-0632-3. Epub 2018 Nov 2. PMID 30386949